CLINICAL TRIAL: NCT01841853
Title: Livslots Angered - A Randomized Controlled Trial of a Community-based Health-promoting and Disease-preventive Program for Older Foreign Born Adults
Brief Title: RCT of Health-promoting Intervention for Older Foreign-born Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Livslots Angered
Record Dates: First submitted 2013-04-10; First posted 2013-04-29 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Health Behavior
Keywords: Elderly; Health promotion; Randomized controlled study; Immigrant; Vulnerable population; ADL; KASAM; Implementation
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Senior meetings (Experimental): The intervention will comprise four weekly meetings in small groups (4-6 participants) in addition to an individual follow-up home visit two to three weeks after the last senior meeting.The main purpose of the senior meetings is to give information and facilitate discussion of the ageing process and provide tools and suggest strategies to enable the clients to solve the various problems that may arise at home in order to remain living at home in a safe and secure way. The information will also include what the municipality provides in the form of local meeting places, activities run by local associations, physical training for seniors, walking groups, possibilities of offering or accepting help on a voluntary basis. Furthermore, they will be informed about help and support available in their city district. Identification of risks for, and advice on, how to prevent falls will also be included.
  Interventions: Behavioral: Senior meetings
- Control group (No Intervention): The control group will receive conventional care on their own initiative.

INTERVENTIONS:
Behavioral: Senior meetings — The intervention will be led by professionals such as a registered occupational therapist, a nurse, a physical therapist, and a social worker. The intervention will comprise four weekly meetings in small groups (4-6 participants) in addition to an individual follow-up home visit two to three weeks after the last senior meeting. To use groups involve the possibility of peer education where participants in a person-centeredness perspective are seen as experts on their own situation and learn from each other. The relationship between the personnel and the participants in the senior meetings can be described as a partnership. Respect for the participant and his/her values, and that the participant gets an opportunity to maintain and develop their own power over their own everyday activities will be essential in the meeting.
  Arms: Senior meetings

SUMMARY:
The overarching aim with this study was to develop, implement and evaluate a health promoting programme for people from Finland or the Western Balkan region, who were 70 years of age or older and independent daily activites (1). The aim of the programme was to prevent or delay dependence in daily activities, health decline, and frailty. The study focused on both evaluation and implementation and the data collection finished in 2016

DETAILED DESCRIPTION:
The study has developed tools for collaboration between the target group, staff and researchers, as well as with tools to bridge barriers to health promotion. For example, alternative ways to recruit participants and to collect and analyse data in studies with and for people who are ageing in a migration context.

The findings describe how a person-centred approach could be used to make use of the resources of the target groups, and visualise methods to bridge linguistic barriers. The education material from Older people in the risk zone has also been translated to Bosnian Serbo-Croatian and Finnish.

ELIGIBILITY:
Inclusion Criteria:

* Foreign-born from Finland or any of five countries in the Western Balkans (Bosnia-Herzegovina, Croatia, Macedonia, Montenegro, and Serbia)
* 70 years of age or older
* Living in Angered, Gothenburg
* Living in their ordinary housing
* Not dependent on informal or formal help in daily activities

Exclusion Criteria:

* Impaired cognition, Mini Mental State Examination (MMSE) below 80% of administered items

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 131 (Actual)
Dates: Start 2012-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change of Activities of Daily Life (ADL) | change from baseline at 6 months and 1 year
  The ADL-staircase
Change of Sense of Coherence (KASAM) | change from basline at 6 months and 1 year
  KASAM (by Antonovsky)

SECONDARY OUTCOMES:
Change of Fatigue | baseline, 6 months, and 1 year
  The Mob-T scale
Change of Grip strength | baseline, 6 months, and 1 year
  North Coast-dynamometer
Change of Physical activity | basline, 6 months, and 1 year
  Questionnaire and Physical and domestic activity scale
Change of Balance | basline, 6 months, and 1 year
  The balance scale
Change of Gait speed | basline, 6 months, and 1 year
  Four-meter walking test
Change of Weight loss | basline, 6 months, and 1 year
  The Göteborg Quality of Life Instrument
Change of Cognition | basline, 6 months, and 1 year
  Mini Mental State Examination (MMSE)
Change of Visual impairment | basline, 6 months, and 1 year
  KM-visual acuity chart
Change of Falls | basline, 6 months, and 1 year
  Questionnaire
Change of Fear of falls | baseline, 6 months, 1 year
  FES-I
Change of Illness | Baline, 6 months, and 1 year
  CIRS-G
Change of Symptoms | Basline, 6 months, and 1 year
  The Göteborg Quality of Life Instrument
Change of Change of Depression | Baseline, 6 months, and 1 year
  GDS 20
Health-care consumption | Baseline, 6 months, and 1 year
  Register data

CONTACTS AND LOCATIONS:
Overall Officials: Synneve Dahlin-Ivanoff, Professor, Study Director — Göteborg University
Locations (1):
- Synneve Dahlin-Ivanoff, Gothenburg, Sweden

REFERENCES:
- [Derived] Gustafsson S, Lood Q, Wilhelmson K, Haggblom-Kronlof G, Landahl S, Dahlin-Ivanoff S. A person-centred approach to health promotion for persons 70+ who have migrated to Sweden: promoting aging migrants' capabilities implementation and RCT study protocol. BMC Geriatr. 2015 Feb 14;15:10. doi: 10.1186/s12877-015-0005-4. PMID 25887506
- [Derived] Lood Q, Gustafsson S, Dahlin Ivanoff S. Bridging barriers to health promotion: a feasibility pilot study of the 'Promoting Aging Migrants' Capabilities study'. J Eval Clin Pract. 2015 Aug;21(4):604-13. doi: 10.1111/jep.12345. Epub 2015 Mar 23. PMID 25810033